CLINICAL TRIAL: NCT06947941
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Safety and Efficacy of KarXT + KarX-EC for the Treatment of Psychosis Associated With Alzheimer's Disease
Brief Title: A Study to Evaluate Safety and Efficacy of KarXT + KarX-EC as a Treatment for Psychosis Associated With Alzheimer's Disease (ADEPT-5)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN012-0034
Record Dates: First submitted 2025-04-25; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease; Psychosis
Keywords: Alzheimer disease; Alzheimer; Dementia; Psychosis
MeSH Terms: conditions — Alzheimer Disease; Psychotic Disorders; Dementia | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: KarXT + KarX-EC Arm Matching Placebo
- KarXT + KarX-EC Arm (Experimental)
  Interventions: Drug: KarXT; Drug: KarX-EC

INTERVENTIONS:
Drug: KarXT — Specified dose on specified days
  Other Names: BMS-986510; Xanomeline/Trospium Chloride
  Arms: KarXT + KarX-EC Arm
Drug: KarX-EC — Specified dose on specified days
  Other Names: BMS-986519; Xanomeline Enteric-coated
  Arms: KarXT + KarX-EC Arm
Drug: KarXT + KarX-EC Arm Matching Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate KarXT + KarX-EC as a treatment for psychosis associated with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 55 to 90 years of age, inclusive, at the time of Screening (Visit 1).
* Participants must be diagnosed with Alzheimer's disease in accordance with the 2024 NIA-AA criteria.
* Participants must have a magnetic resonance imaging (MRI) or computed tomography (CT) scan of the brain (completed within the past 5 years) taken during or subsequent to the onset of dementia to rule out other central nervous system (CNS) disease that could account for the dementia syndrome, eg, major stroke, neoplasm, subdural hematoma.
* Participants must have a history of psychotic symptoms (meeting International Psychogeriatric Association criteria) for at least 2 months prior to Screening (Visit 1) (participants may or may not have symptoms of agitation).

Exclusion Criteria:

* Participants must not have psychotic symptoms that are primarily attributable to a condition other than the AD causing the dementia, eg, schizophrenia, schizoaffective disorder, delusional disorder, or mood disorder with psychotic features.
* Participants must not have history of major depressive episode with psychotic features during the 12 months prior to Screening, or history of bipolar disorder, schizophrenia, or schizoaffective disorder.
* Participants must not have certain safety concerns, including certain laboratory test irregularities.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1046 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2027-09-27 (Estimated); Study Completion 2027-10-25 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Neuropsychiatric Inventory-Clinician: Hallucinations and Delusions (NPI-C: H+D) Score | Up to Week 12

SECONDARY OUTCOMES:
Change From Baseline in Clinical Global Impressions-Severity (CGI-S) Score | Up to Week 12
Change From Baseline in Neuropsychiatric Inventory-Clinician Rating Scale (NPI-C) Core Score | Up to Week 12
  NPI-C Core Score includes assessment for hallucinations, delusions, agitation, and aggression domains
Change From Baseline in NPI-C: Agitation Score | Up to Week 12
Change From Baseline in NPI-C Core Score: Caregiver Distress Scale | Up to Week 12
  NPI-C Core Score: Caregiver Distress Scale includes assessment for hallucinations, delusions, agitation, and aggression domains
Responder Rate | Up to Week 12
  Responder rate is defined as improvement from baseline in NPI-C: H+D score ≥ 40% by the end of Week 12
Change From Baseline in Cohen-Mansfield Agitation Inventory International Psychogeriatric Association (CMAI-IPA) Score | Up to Week 12
Change From Baseline in CMAI Total Score | Up to Week 12
Number of Participants With Adverse Events (AEs) | Up to approximately Week 18
Number of Participants With Serious Adverse Events (SAEs) | Up to approximately Week 18
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to approximately Week 18
Number of Participants With TEAEs Leading to Discontinuation | Up to approximately Week 18
Number of Participants With Spontaneously Reported Procholinergic Symptoms | Up to approximately Week 18
  Procholinergic symptoms include nausea, vomiting, and diarrhea.
Number of Participants With Spontaneously Reported Anticholinergic Symptoms | Up to approximately Week 18
  Anticholinergic symptoms include dry mouth, constipation, urinary retention and blurred vision.
Number of Participants With AEs of Special Interest (AESIs) That Require Drug-induced Liver Injury (DILI) Monitoring | Up to approximately Week 18
  AESIs requiring DILI monitoring such as symptomatic orthostasis, syncope, and elevated liver enzymes will be evaluated.
Change From Baseline in Barnes Akathisia Rating Scale (BARS) Score | Up to approximately Week 14
Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Score | Up to approximately Week 14
Change From Baseline in International Prostate Symptom Score (IPSS) | Up to approximately Week 14
  This will be measured in males only.
Change From Baseline in Body Weight | Up to approximately Week 14
Change From Baseline in Body Mass Index (BMI) | Up to approximately Week 14
Number of Participants With Clinically Significant Changes in Orthostatic Vital Sign: Heart Rate (HR) | Up to approximately Week 14
  This includes measuring of HR, both supine and standing or seated and upon standing after 2 minutes.
Number of Participants With Clinically Significant Changes in Orthostatic Vital Sign: Blood Pressure (BP) | Up to approximately Week 14
  This includes measuring of systolic and diastolic BP, both supine and standing or seated and upon standing after 2 minutes.
Number of Participants With Clinically Significant Changes in Laboratory Evaluations: Hematology | Up to approximately Week 14
Number of Participants With Clinically Significant Changes in Laboratory Evaluations: Clinical Chemistry | Up to approximately Week 14
Number of Participants With Clinically Significant Changes in Laboratory Evaluations: Coagulation Parameters | Up to approximately Week 14
Number of Participants With Clinically Significant Changes in Laboratory Evaluations: Prolactin Levels | Up to approximately Week 14
Number of Participants With Clinically Significant Changes in Laboratory Evaluations: Urinalysis | Up to approximately Week 14
Number of Participants With Clinically Significant Changes in Laboratory Evaluations: Drug Screening | Up to approximately Week 14
Number of Participants With Clinically Significant Changes in 12-lead Electrocardiogram (ECG) | Up to approximately Week 14
Number of Participants With Suicidal Ideations and Behavior as Assessed Using the Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to approximately Week 18
Number of Participants With Cognitive Impairment as Assessed by Mini-mental State Examination (MMSE) | Up to approximately Week 14
Number of Participants With Cognitive Impairment as Assessed by 13-item Variation of ADAS-Cog Scale (ADAS-Cog-13) | Up to approximately Week 14

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com